CLINICAL TRIAL: NCT05076188
Title: PARamedical Abnormalties Detection of Traumatic Bone Lesion of the extremitIeS
Acronym: PARADIS_1
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Paradis_1
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-03

CONDITIONS: Radiography; Emergencies; Diagnostic
MeSH Terms: conditions — Emergencies; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Emergency radiography — The intervention is to determine how the radiographer classify emergency radiography.

SUMMARY:
This study assesses the performance of radiographers in detecting radiological anomalies of the appendicular skeleton in emergency department. This is a retrospective study comparing the radiographers' diagnostic performance before and after dedicated training, assisted or not by artificial intelligence software. All performances will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Working in an emergency radiography department Volunteer to participate in the study

Exclusion Criteria:

* Planned departure from the establishment within 12 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Radiographer : a health practionner with official autorisation to use X-ray imagery.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the radiographers' diagnostic performance to issue an advisory opinion to X-ray reading of the appendicular skeleton in emergency department | 2 hours
  The primary outcome measure evaluation radiographers' diagnostic will use accurancy, sensibility and specificity.

SECONDARY OUTCOMES:
Quantify the proportion of radiographers reaching the goal of 90% accurancy | 4 months
  This is a proportion in % of performance radiographers' diagnosctic treshold
Quantify and qualify Radiographers diagnostic changes before and after the in house training. | 4 months
  This a proportion in % about the progression of performance radiographers'diagnostic in the formation.
Evaluate the performance of the association of AI and radiographer after training | 4 months
  Thiis output is the difference between accurancy, sensibility and sensitivity with or without IA.

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. de Poitiers, Poitiers, France